CLINICAL TRIAL: NCT02846090
Title: Dexmedetomidine as an Additive to Local Anaesthesia to Decrease Intraocular Pressure in Glaucoma Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, Hassan Mohamed Ali, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01001733687
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- D50 Dexmedetomidine 50 micrograms group (Experimental): peribulbar block was given using 10 ml of a mixture of local anesthetics. The mixture was composed of 5 ml of 0.5% bupivacaine +4.5 ml of 2% lidocaine +0.5ml of 50 micrograms of Dexmedetomidine with 150 IU hyaluronidase.
  Interventions: Drug: Dexmedetomidine to reduce the IOP
- D25 Dexmedetomidine 25 micrograms group (Experimental): peribulbar block was given using 10 ml of a mixture of local anesthetics. The mixture was composed of 5 ml of 0.5% bupivacaine + 4.5 ml of 2% lidocaine +0.5ml of 25 micrograms of Dexmedetomidine with 150 IU hyaluronidase.
  Interventions: Drug: Dexmedetomidine to reduce the IOP
- control (Placebo Comparator): peribulbar block was given using 10 ml of a mixture of local anesthetics without Dexmedetomidine. The mixture was composed of 5 ml of 0.5% bupivacaine +4.5 ml of 2% lidocaine +0.5ml with 150 IU hyaluronidase.
  Interventions: Drug: Dexmedetomidine to reduce the IOP

INTERVENTIONS:
Drug: Dexmedetomidine to reduce the IOP — Dexmedetomidine 50 micrograms group (D50) in which peribulbar block was given using 10 ml of a mixture of local anesthetics. The mixture was composed of 5 ml of 0.5% bupivacaine +4.5 ml of 2% lidocaine +0.5ml of 50 micrograms of Dexmedetomidine with 150 IU hyaluronidase.
  Other Names: reduction of OCULAR HYPERTENSION

SUMMARY:
Nowadays, a number of cases with increased intraocular pressure and glaucoma have been shown a huge increase . This is because of the increase the geriatric population in the community and advanced medical care. Surgical correction, as a treatment, solves this problem greatly especially with the modern surgical techniques .

Peribulbar block reduced the admission discharge time and reduced the burden on both the patients and the medical team. On the other hand, it carries the risk of increased intraocular pressure (IOP). Which, subsequently, limit its usage in glaucoma surgery.

Dexmedetomidine, as an alpha 2 agonist, has a well-established role in decreasing intraocular pressure (IOP). This effect has been shown at a histological level and clinical level

DETAILED DESCRIPTION:
Nowadays, number of cases with increased intraocular pressure and glaucoma has been shown a huge increase . This is because of the increase the geriatric population in the community and advanced medical care. Surgical correction, as a treatment, solves this problem greatly especially with the modern surgical techniques .

Peribulbar block reduced the admission discharge time and reduced the burden on both the patients and the medical team. On the other hand, it carries the risk of increased intraocular pressure (IOP). Which, subsequently, limit its usage in glaucoma surgery .

Dexmedetomidine, as an alpha 2 agonist, has a well established role in decreasing intraocular pressure (IOP). This effect has been shown at a histological level and clinical level . It has been tested in many studies before as an additive to local anaesthetic to augment the effect of the block and to achieve an accepted level of patient sedation (**). Many routes have been tested such as intravenous infusion, intramuscular injection and topically with the local anaesthesia . There is a debate about the best route and the optimum dose that can achieve the desired clinical effect with the least side effects.

There is no study, till now, has examined the effect of Dexmedetomidine in a diseased eye with pathology that leads to increased IOP. This study states the hypothesis that Dexmedetomidine locally as an additive to local anaesthesia in different doses, not only will increase the duration of the block or achieve some level of sedation, but also can reduce the IOP in this diseased eye to a level that will help the surgical conditions and improve the surgical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Any patients who were ASA I-III, age more than 25 and less than 80 with diagnosed increased intraocular pressure and were legible for surgical correction

Exclusion Criteria:

* Patients with known allergy to the medications to be given, ASA more than III, age less than 25 or more than 80, dementia, deafness, psychological disease, difficult to communicate, cannot lay flat, INR more than 1.7 or with significant coagulopathy

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
IOP before the block, after the message and before the surgical incision, after the end of the surgery | one hour
  IOP before the block, after the message and before the surgical incision, after the end of the surgery

SECONDARY OUTCOMES:
Onset of the block | 2 min
  the time elapsed between the end of the block and the complete anaesthesia and complete or partial akainesia

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided